CLINICAL TRIAL: NCT01418222
Title: Randomized, Double-Blind, Phase II Study of FOLFOX/Bevacizumab With Onartuzumab (MetMAb) Versus Placebo as First-Line Treatment for Patients With Metastatic Colorectal Cancer
Brief Title: FOLFOX/Bevacizumab With Onartuzumab (MetMAb) Versus Placebo as First-Line Treatment in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: SCRI Development Innovations, LLC (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO27827
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Folfox protocol; Bevacizumab; Leucovorin; onartuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: 5-FU; Drug: FOLFOX regimen; Drug: bevacizumab [Avastin]; Drug: leucovorin; Drug: onartuzumab [MetMAb]
- B (Active Comparator)
  Interventions: Drug: 5-FU; Drug: FOLFOX regimen; Drug: Placebo; Drug: bevacizumab [Avastin]; Drug: leucovorin

INTERVENTIONS:
Drug: 5-FU — Intravenous repeating dose
Drug: FOLFOX regimen — Intravenous repeating dose
Drug: Placebo — Intravenous repeating dose
  Arms: B
Drug: bevacizumab [Avastin] — Intravenous repeating dose
Drug: leucovorin — Intravenous repeating dose
Drug: onartuzumab [MetMAb] — Intravenous repeating dose
  Arms: A

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of FOLFOX/bevacizumab with onartuzumab (MetMAb) versus placebo as first-line treatment in patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum in patients with metastatic (Stage IV) disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Measurable disease by RECIST criteria
* Adequate organ system function, as defined by protocol

Exclusion Criteria:

* Prior systemic or radiation therapy for metastatic colorectal cancer
* Adjuvant chemotherapy (and/or chemoradiation) for colorectal cancer within 12 months prior to date of diagnosis of metastatic disease
* Previously untreated brain metastases
* History of hypersensitivity to active or inactive excipients of any component of treatment, or known dipyrimidine dehydrogenase deficiency
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* History of hematemesis or hemoptysis </= 1 months prior to study enrollment
* Significant cardiovascular disease or disorder
* History of abdominal fistula or gastrointestinal perforation </= 6 months prior to Day 1
* Positive for hepatitis B, hepatitis C or HIV infection
* Other active cancers or history of treatment for invasive cancer within the last 5 years, except for non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2011-09-14 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

PRIMARY OUTCOMES:
Progression-free survival: time from randomization to tumor progression or death, tumor assessments according to RECIST criteria | up to 4 years

SECONDARY OUTCOMES:
Response rate (complete response + partial response) | up to 4 years
Time to treatment failure: from randomization to treatment discontinuation for any reason including disease progression, treatment toxicity, and death | up to 4 years
Overall survival | up to 4 years
Safety: Incidence of adverse events | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (23):
- United States (23):
  - Almac Clinical Technologies, San Francisco, California
  - Rocky Mountain Cancer Centers; Bone and Marrow Trans, Denver, Colorado
  - Florida Cancer Specialists; SCRI, Fort Myers, Florida
  - Florida Hospital Cancer Inst, Orlando, Florida
  - Georgia Cancer Specialists - Northside, Atlanta, Georgia
  - University of Chicago; Hematology/Oncology, Chicago, Illinois
  - Ingalls Cancer Research Center, Harvey, Illinois
  - Ingalls Memorial Hospital; Cancer Research Center, Harvey, Illinois
  - Baptist Hospital East, Louisville, Kentucky
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Saint Louis Cancer Care, LLP, Bridgeton, Missouri
  - Research Medical Center - Antibiotic Research Associates, Inc., Kansas City, Missouri
  - Hem-Onc Assoc of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Toledo Comm. Onc. Program, Toledo, Ohio
  - University of Oklahoma; Stephenson Oklahoma Canc Ctr, Oklahoma City, Oklahoma
  - South Carolina Oncology Associates - SCRI, Columbia, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Tennessee Onc., PLLC - SCRI, Nashville, Tennessee
  - Ctr for Cancer and Blood Disorders, Fort Worth, Texas
  - South Texas Oncology & Hematology, P.A., San Antonio, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Derived] Bendell JC, Hochster H, Hart LL, Firdaus I, Mace JR, McFarlane JJ, Kozloff M, Catenacci D, Hsu JJ, Hack SP, Shames DS, Phan SC, Koeppen H, Cohn AL. A Phase II Randomized Trial (GO27827) of First-Line FOLFOX Plus Bevacizumab with or Without the MET Inhibitor Onartuzumab in Patients with Metastatic Colorectal Cancer. Oncologist. 2017 Mar;22(3):264-271. doi: 10.1634/theoncologist.2016-0223. Epub 2017 Feb 16. PMID 28209746